CLINICAL TRIAL: NCT06494293
Title: How Many Patients Suffering Major Trauma Would be Eligible for a Pre-hospital Transfusion: A Multicentre Retrospective Study.
Brief Title: How Many Patients Suffering Major Trauma Would be Eligible for a Pre-hospital Transfusion
Acronym: TRAP
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Collaborators: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1024
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Trauma Injury
Keywords: Major trauma; Mobile Intensive Care Unit (MCIU); Out of hospital emergency care; Blood transfusion
MeSH Terms: conditions — Accidental Injuries | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data collection: Collection of medical data from MICU intervention file and patient medical files from participating centres
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Collection of medical data from MICU intervention file and patient medical files from participating centres

SUMMARY:
The aim of the study is to measure the number of patients being cared for by a medical team for major trauma who could benefit from a transfusion labile blood products and thus provide a scientific argument in favour of supplying labile blood products to pre-hospital

DETAILED DESCRIPTION:
In France, pre-hospital resuscitation of major trauma patients does not use labile blood products, except in exceptional circumstances. The physician staffed Mobile Intensive Care Unit (MICU) are not equipped with this type of product. The first cause of death compatible with survival in the event of pre-hospital treatment identified in major trauma in war medicine is exsanguination. Mortality in haemorrhagic shock occurs rapidly and appears to be significantly reduced if transfusions are performed early. Early transfusion has proved its worth in the military context, leading the armed forces health service to recommend transfusion as a first-line treatment as quickly as possible, from the moment the patient is taken into care on the battlefield. More recently, in the North American civilian pre-hospital setting, the PAMPer study included 501 patients, 230 of whom were transfused with fresh frozen plasma (FFP - 2 units). The authors reported a significant reduction in mortality at D+30 in the FFP group (23.2% vs 33%; p=0.03). It therefore seems that transfusion as early as possible is associated with a reduction in mortality in the context of major trauma.

The aim of the study is to measure the number of patients being cared for by a medical team for major trauma who could benefit from a transfusion labile blood products and thus provide a scientific argument in favour of supplying labile blood products to pre-hospital.

ELIGIBILITY:
Inclusion Criteria :

* Patients over 18
* Taken care of by a MICU team from participating centres
* Victims of major trauma requiring transport to an emergency/recovery unit or declared dead during care
* Informed and did not object to the collection of his data for research purposes during his lifetime

Exclusion Criteria :

* Traumatological reason for departure not confirmed in the emergency medical services report
* Patient care of by the MICU for secondary transport (transport from one hospital to another)
* Patient died without resuscitation by a professional
* Patient with manifest isolated closed head injury
* Patient deprived of civil rights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being cared for by a medical team for major trauma requiring transport to an emergency/recovery unit or declared dead during care between the 1st January 2023 and the 31th December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of the proportion of patients being cared for a medical team for major trauma who could have benefited from a pre-hospital transfusion | At the end of the study, an average of 4 month
  The main analysis criterion will be the presence, during pre-hospital management, of a massive and immediate blood transfusion criterion measured by the ABC (Assessment of Blood Consumption) score between the arrival of the MICU and 10 minutes before arrival at the hospital.
  This score is used to predict the need for massive transfusion, defined in particular as the administration of 4 labile blood products within the first hour of hospital care.
  This score will be calculated retrospectively on the basis of data collected from the medical record at the time the patient is taken into medical care, and then every 10 minutes during the course of the care until 10 minutes after arrival at hospital.
  An ABC score greater than or equal to 2 indicates a probability of massive transfusion greater than 75%. We will consider a score >= 2 as "probably requiring a pre-hospital transfusion".

SECONDARY OUTCOMES:
Evaluation of the concordance between the number of patients who received a transfusion during their pre-hospital care and the ABC (Assessment of Blood Consumption) score | At the end of the study, an average of 4 month
  The concordance will be assessed by the presence of at least one transfusion, whatever the volume between the work-up and arrival at hospital.
Assessment of patient mortality on arrival at the resuscitation/recovery centre | At the end of the study, an average of 4 month
  Mortality will be assessed by the number of patients alive on arrival of the MICU and dead on arrival at hospital.
Assessment of patients care time | At the end of the study, an average of 4 month
  Care time will be determined by the time between the arrival of the medical team and arrival at the hospital.
Assessment of the number of patients who could have benefited of a REBOA (Resuscitative Endovascular Balloon Occlusion of the Aorta) | At the end of the study, an average of 4 month
  This number will be assessed as follow : number of patients potentially eligible for placement of a REBOA in terms of the presence of abdominal or pelvic bleeding on ultrasound, a PAS > 90 mmHg despite 3 mg/h NAD (noradrenaline) and the absence of thoracic trauma or Supra Aortic Trunks (SATs).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Dorian WOLFF, Principal Investigator — Hôpital NOVO
Locations (4):
- France (4):
  - Resuscitation Services (SMUR) Ballanger - Centre Hospitalier Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Resuscitation Services (SAMU/SMUR) - Hôpital NOVO -Beaumont/Oise Site, Beaumont-sur-Oise
  - Resuscitation Services (SAMU/SMUR) - Hôpital NOVO -Pontoise Site, Pontoise
  - Resuscitation Services (SMUR) Delafontaine - Centre Hospitalier de Saint-Denis, Saint-Denis

REFERENCES:
- [Background] Bichot A, Pasquier P, Martinaud C, Corcostegui SP, Boutot F, Cazes N, Boutillier du Retail C, Travers S, Galant J. Use of prehospital transfusion by French emergency medical services: A national survey. Transfusion. 2023 May;63 Suppl 3:S241-S248. doi: 10.1111/trf.17374. Epub 2023 Apr 20. PMID 37071770
- [Background] Vitalis V, Carfantan C, Montcriol A, Peyrefitte S, Luft A, Pouget T, Sailliol A, Ausset S, Meaudre E, Bordes J. Early transfusion on battlefield before admission to role 2: A preliminary observational study during "Barkhane" operation in Sahel. Injury. 2018 May;49(5):903-910. doi: 10.1016/j.injury.2017.11.029. Epub 2017 Nov 23. PMID 29248187
- [Background] Sperry JL, Guyette FX, Brown JB, Yazer MH, Triulzi DJ, Early-Young BJ, Adams PW, Daley BJ, Miller RS, Harbrecht BG, Claridge JA, Phelan HA, Witham WR, Putnam AT, Duane TM, Alarcon LH, Callaway CW, Zuckerbraun BS, Neal MD, Rosengart MR, Forsythe RM, Billiar TR, Yealy DM, Peitzman AB, Zenati MS; PAMPer Study Group. Prehospital Plasma during Air Medical Transport in Trauma Patients at Risk for Hemorrhagic Shock. N Engl J Med. 2018 Jul 26;379(4):315-326. doi: 10.1056/NEJMoa1802345. PMID 30044935
- [Background] Eastridge BJ, Mabry RL, Seguin P, Cantrell J, Tops T, Uribe P, Mallett O, Zubko T, Oetjen-Gerdes L, Rasmussen TE, Butler FK, Kotwal RS, Holcomb JB, Wade C, Champion H, Lawnick M, Moores L, Blackbourne LH. Death on the battlefield (2001-2011): implications for the future of combat casualty care. J Trauma Acute Care Surg. 2012 Dec;73(6 Suppl 5):S431-7. doi: 10.1097/TA.0b013e3182755dcc. PMID 23192066
- [Background] Fox EE, Holcomb JB, Wade CE, Bulger EM, Tilley BC; PROPPR Study Group. Earlier Endpoints are Required for Hemorrhagic Shock Trials Among Severely Injured Patients. Shock. 2017 May;47(5):567-573. doi: 10.1097/SHK.0000000000000788. PMID 28207628